CLINICAL TRIAL: NCT01896986
Title: HPV Immunisation Protecting Special Risk Group Patients From Cervical Cancer: 5 Year Follow-up Post-vaccination
Brief Title: HPV Vaccination in Special Risk Groups: 5 Year Follow-up
Status: Terminated | Type: Observational
Why Stopped: recruitment problems
Sponsor: Murdoch Childrens Research Institute (Other)
Collaborators: Monash Medical Centre (Other)
Responsible Party: Principal Investigator, Nigel Crawford, Medical Head Immunisation, General Paediatrician, Murdoch Childrens Research Institute
Other Study IDs: HPV girls 5year followup
Record Dates: First submitted 2013-06-25; First posted 2013-07-11 (Estimated); Results first posted 2017-06-15 (Actual); Last update posted 2017-06-15 (Actual); Status verified 2017-03

CONDITIONS: PRD (Paediatric Rheumatological Disease); IBD (Inflammatory Bowel Disease)
Keywords: Special risk patients; Immunosuppressive biologic treatments; PRD (Paediatric Rheumatological Disease); IBD (Inflammatory Bowel Disease)
MeSH Terms: conditions — Inflammatory Bowel Diseases

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (2):
- PRD patrients: Children/adolescent females 12-26 years with a PRD such as JIA (Juvenile Idiopathic Arthritis) or SLE (Systemic Lupus Erythematosus)
  Subgroups:
  1. receiving immunosuppressant therapy
  2. not on immunosuppressant therapy
- IBD patients: Children/adolescent females 12-26 years diagnosed with IBD.
  Subgroups:
  3. receiving immunosuppressant therapy 4. not on immunosuppressant therapy

SUMMARY:
In 2007-2009 the investigators conducted a study to determine the immunogenicity response to HPV vaccine in special risk patients known to be at increased risk of abnormal cervical cytology. The serological response to the vaccine was measured 1 month post the third and final dose (n=70) finding a robust response overall.

The aim of this follow-on study is to provide data on the long-term protection offered by the HPV vaccination. The persistence of antibody 5 years post immunisation is unknown and the impact on cervical cytology abnormalities in these special risk groups is important.

The study results will help inform national immunisation program recommendations re- booster HPV vaccine doses.

DETAILED DESCRIPTION:
This study is an open interventional study based at two paediatric tertiary centres in Melbourne, Australia. It is specifically looking at the long term immunogenic response to the 4 valent HPV vaccine (4vHPV) Gardasil in paediatric rheumatology disease (PRD) and Irritable bowel disease (IBD) in participants who complete the primary HPV immunological study.

The study participant's response to the vaccine will be compared to Merck historical age-matched controls as there is currently no serological correlate of protection for the HPV vaccine.

The participants have already received the vaccine as part of the Australian federally funded catch up program which will run until mid-2009. All participants are part of 'Special risk groups'; which as defined by the Australian Immunisation Handbook, as patients who may have:

1. special vaccination needs (e.g. children/ adolescents with a chronic medical condition) ; or
2. a suboptimal response to vaccination (e.g. due to impaired immunity); or
3. an increased risk of adverse events following immunization (AEFI)

The 'special risk groups' currently included in the study are:

1. PRD- Paediatric Rheumatological Diseases
2. IBD- Inflammatory Bowel Disease

Number of participants

Total number of patients to be recruited is N = 60

The aim is to recruit n= 45 patients from PRD and n=15 patients from IBD.

Immunisation history will be correlated with the HPV register.

Main outcome measures

The primary immunogenicity endpoint will be serum antibody by month 60 (i.e. 5 years post 3rd and final dose of 4vHPV vaccine).

Antibody titres are determined by using type-specific competitive neutralising antibody to epitopes on virus like particles (VLP). This will be for each of the 4 serotypes in the vaccine [6,11,16,18], with geometric mean titre (GMT) will be measured in mMU; and will be compared with GMT from historical age-matched controls.

Frequency of assessment

There will only be one immunogenicity assessment point, 60 month post the third and final dose of 4vHPV vaccine.

Primary Objective:

• Long term immunogenicity of the quadrivalent 4/6/11/18 HPV vaccine Gardasil® by following up a cohort of adolescent females aged 16-30 years with PRD or IBD, 5 years post HPV vaccination at the Royal Children's Hospital (RCH) Melbourne. Antibody titres are determined by using type specific neutralizing antibody.The geometric mean titre (GMT) will be measured in mMU; with a type specific cutoff for the assay (> 20mMU/ml for the HPV6; > 16mMU/ml for the HPV11; > 20mMU/ml for the HPV16 and >24mMU/ml for the HPV18). [13,15] HPV serology will be performed using competitive Luminex based immunoassays.

Secondary Objective:

• The safety of the HPV vaccine in the 2 (PRD, IBD) study groups, measured by the number of adverse events reported by study participants.

ELIGIBILITY:
Inclusion Criteria:

* Females who participated in the initial HPV vaccine immunogenicity study in 2007.

Exclusion Criteria:

* Inability to provide informed consent

Ages: 12 Years to 26 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Child, Adult
Study Population: In 2007 we began a clinical audit of the 'special risk patients' within two subgroups (PRD&IBD). From April 2007- March 2010 there were 64 special risk female participants including 38 PRD patients of which 28 had juvenile idiopathic arthritis (JIA). The other subgroups included: 14 IBD; 10 paediatric cancer; 1 SOTR (solid organ transplant recipient) and 1 CRD (Chronic Renal Disease). The median age at the first dose of 4vHPV vaccine administration was 14.7 years [range 11.8 to 24.7].
  The overall results were good with all participants showing at least some level of antibody protection against HPV.
  Long-term follow-up will help determine the requirement for booster vaccine doses, including those patients treated with combination immunosuppressive therapies.
Sampling Method: Non-Probability Sample
Enrollment: 37 (Actual)
Dates: Start 2012-03; Primary Completion 2012-03 (Actual); Study Completion 2012-03 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Nigel Crawford, PhDMPHMBBS, Principal Investigator — Royal Childrens Hospital
Locations (1):
- Royal Childrens Hospital, Melbourne, Victoria, Australia

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | PRD Patrients | IBD Patients
Started | 14 | 23
Completed | 0 | 0
Not Completed | 14 | 23
Not completed — samples lost | 14 | 23

BASELINE CHARACTERISTICS:
Population: Group A:PRD - Children/adolescent females 12-26 years with a PRD such as JIA (Juvenile Idiopathic Arthritis) or SLE (Systemic Lupus Erythematosus) Group B: IBD (Inflammatory Bowel Disease) Children/adolescent females 12-26 years diagnosed with IBD.
Groups:
- Total: Total of all reporting groups
Arm/Group | PRD Patrients | IBD Patients | Total
Number analyzed (Participants) | 14 | 23 | 37
Age, Continuous [Mean (Full Range); unit: years] | 19 [17 to 24] | 23 [12 to 30] | 21 [12 to 30]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 14 | 23 | 37
  Male | 0 | 0 | 0
Region of Enrollment [Number; unit: participants]
  Australia | 14 | 23 | 37

OUTCOME MEASURES:

1. Primary Outcome: Immunogenicity to HPV Vaccine Gardasil
Description: To evaluate the long term immunogenicity of the quadrivalent 4/6/11/18 HPV vaccine Gardasil® by following up a cohort of adolescent females aged 16-30 years with PRD or IBD, 5 years post HPV vaccination at the Royal Children's Hospital (RCH) Melbourne .
Time Frame: 12 months
Population: No immunogenicity data collected as samples were lost.
Groups:
- PRD Patrients: Children/adolescent females 12-26 years with a PRD such as JIA (Juvenile Idiopathic Arthritis) or SLE (Systemic Lupus Erythematosus)
  Subgroups:
  1. receiving immunosuppressant therapy
  2. not on immunosuppressant therapy
  No samples analysed.
- IBD Patients: Children/adolescent females 12-26 years diagnosed with IBD.
  Subgroups:
  3. receiving immunosuppressant therapy 4. not on immunosuppressant therapy
  No samples analysed.
Arm/Group | PRD Patrients | IBD Patients
Number analyzed (Participants) | 0 | 0
Value | 0 | 0

ADVERSE EVENTS:
Time Frame: No drugs were given to patient population so adverse event reporting was not applicable.
Description: No drugs were given to patient population so adverse event reporting was not applicable.
Groups:
- PRD Patrients: Children/adolescent females 12-26 years with a PRD such as JIA (Juvenile Idiopathic Arthritis) or SLE (Systemic Lupus Erythematosus)
  Subgroups:
  1. receiving immunosuppressant therapy
  2. not on immunosuppressant therapy
  no adverse events
- IBD Patients: Children/adolescent females 12-26 years diagnosed with IBD.
  Subgroups:
  3. receiving immunosuppressant therapy 4. not on immunosuppressant therapy
  no adverse events
Arm/Group | PRD Patrients | IBD Patients
Serious Adverse Events (participants affected / at risk) | 0/0 | 0/0
Other Adverse Events (participants affected / at risk) | 0/0 | 0/0

LIMITATIONS AND CAVEATS:
Study serum samples being misplaced so sample testing could not be done. As such we had no choice but to close this study. This was communicated to the enrolled participants and the RCH ethics department.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No